CLINICAL TRIAL: NCT00767091
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicentric Trial
Brief Title: Study of Rivastigmine to Treat Parkinsonian Apathy Without Dementia
Acronym: CHoPA-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-002578-36; 2008/0817 (Other: sponsor)
Record Dates: First submitted 2008-09-01; First posted 2008-10-06 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2009-03

CONDITIONS: Parkinson's Disease; Apathy; no Dementia
Keywords: Parkinson's disease; Apathy; Rivastigmine; transdermal patch; anticholinesterasic; acetylcholine
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — Rivastigmine; Cholinesterase Inhibitors; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Active Comparator): A: transdermal rivastigmine at 4.6 mg per day during one month then 9.5 mg per day during 5 months.
  Interventions: Drug: rivastigmine
- placebo (Placebo Comparator): transdermal patch of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rivastigmine — transdermal patch of rivastigmine of 9.5 mg/day
  Other Names: cholinesterase inhibitors (Exelon)
  Arms: Active treatment
Drug: placebo — transdermal patch of placebo
  Other Names: transdermal patch without active substance
  Arms: placebo

SUMMARY:
Apathy usually refers to a set of behavioural, emotional and cognitive features as a reduced interest and participation in main activities of daily life, a lack of initiative, a trend toward an early withdrawal from started activities, an indifference and a flattening of affect. We have validated a new specific scale (Lille Apathy Rating Scale, LARS) in order to detect and quantify apathy in Parkinson's disease (PD). Apathy was shown to be frequent in PD with a prevalence of 32%. It has suggested that the medial frontal and limbic cholinergic deficits may underlie apathy in neurodegenerative disorders like Alzheimer's disease (AD). Such a hypothesis is supported by recent evidence indicating the beneficial effects of cholinesterase inhibitors on neuropsychiatric symptoms, mainly apathy, in AD patients. As the efficacy of rivastigmine on cognition has also been shown in PD, we aimed to assess with a randomized, double-blind, placebo-controlled, parallel-group, multicenter trial, the efficacy and acceptability of a 6 months treatment with rivastigmine on apathy in 60 patients with PD without dementia. The primary end point will be the LARS score and the secondary end points will be the cognitive, behavioural and motor symptoms of PD. Two add-on studies will be proposed: first the measure of choline and glutamate peaks on Magnetic Resonance Spectrometry focused on the structures implicated in apathy in order to give insights in the physiopathological mechanisms of the treatment. Secondly, the recording of the REM sleep behavior disorders in relation with the cholinergic part of the pedunculopontine nucleus. Regarding that apathy could be one of the first steps toward PD dementia, treating very early could have substantial implications on the patients and their caregiver.

DETAILED DESCRIPTION:
Overall study duration: 2 years. Planned inclusion period: 12 months. Study duration for individual patients: 7 months (2 weeks between screening and randomization, 6 months of double-blind treatment and then a 2-week wash-out period).

Primary objective (V1 and V6):

To assess efficacy of anticholinesterasic treatment (trans-dermal patch of rivastigmine , Exelon®) on parkinsonian apathy assessed by the Lille Apathy Rating Scale in patients with advanced Parkinson's disease without dementia or depression

Additional Efficacy Endpoints (V1 and V6):

* the NeuroPsychiatric Inventory, the apathy/retardation subscore of the MADRS (tri-dimensional analysis, the Activity of Daily Living scale, the simple and complex reaction times (selective attention), the quality of life (PDQ-39), the "Zarit" scale and the Clinical Global Impression of Change, Independence Scale, Mattis score, MMSE
* Gait: time and number of steps and freezing at the Stand Walk Sit test, the Tinetti scale, the UPDRS I, II, III et IV, the self questionnaire of Giladi
* Sleep quality: during two successive polysomnography recordings (sleep pattern, measures of the rapid eye movement (REM) sleep time, daytime sleepiness (PDSS and Epworth), and Sleep Latency Test
* Magnetic Resonance Spectroscopy on the measures of the choline/creatine and glutamate/creatine peaks (medial frontal cortex, limbic cortex, caudate nucleus, putamen, pedunculopontine nucleus) on 3 Tesla MRI

Safety and Tolerability Endpoints (V1, V3 and V6):

Safety and tolerability will be evaluated with reference to the following:

1. Tolerability :

   Number of subjects (%) who discontinue the study, Number of subjects (%) who discontinue the study due to AEs.
2. Safety Measures :

AE incidence, Safety laboratory values, Vital signs, Blood pressure monitoring, ECG, Physical and neurological examination.

Study Design

Multicentric pilot study: 36-week double blind, placebo-controlled phase. After being found eligible to participate in the study, subjects will be allocated in a 1:1 ratio into one of the following two treatment groups based on a randomization scheme with blocks stratified:

1. one patch of 4.6 mg/day during 1 month, then one patch of 9.5 mg/day during 5 months
2. one patch of placebo during 6 months

Schedule: 7 visits

* Four consultations: screening (V0), randomisation (V1, 15 days after V0), (V3) visit after 3 months and termination (V7, 6 months after randomisation)
* Two phone calls (V2, V4)

Patients :

60 subjects with Parkinson's disease duration of more than 5 years, without dementia (Mattis Dementia Rating Scale ≥ 130, MMSE ≥ 27 and DSM IV), without major depression (MADRS < 18) who have developed apathy (defined by a score of - 16 or more at the LARS) despite an optimal dopaminergic treatment No additional therapy will be permitted during the study.

Investigational Medicinal Product (IMP) & Dosage:

Rivastigmine, or matching placebo, administered by transdermal patch a day in the morning:

4.6 mg a day during one month, 9.5 mg a day during five months

Centres :

Lille :

* Department of Neurology, University Hospital, Lille : Pr L. Defebvre, Pr K. Dujardin, Dr D. Devos, Pr Destee, Mme Delliaux. Dr A Kreisler, Dr C Simonin, Dr C. Moreau
* Department of Pharmacology, Faculté de Médecine, Lille II : R. Bordet
* Department of Clinical Neurophysiology, sleep laboratory : Pr P. Derambure, Dr C. Monaca
* Department of Neuroradiology : Pr J. Pruvo Dr C. Delmaire Dr P. Jissendi, Dr G. Soto Ares, Pr X. Leclerc
* Department of Statistics, CERIM, Faculté de Médecine Lille II : Dr P. Devos, Dr A. Duamel
* Lille III University : Dr P. Sockeel Méthodologiste

Amiens :

- Department of Neurology, University Hospital, Amiens : Pr P. Krystkowiak, Pr O. Godefroy, Dr Gérard, Dr Dupuy, Pr Deramon, Pr JM Macron, Dr Rose

Rouen :

- Department of Neurology, University Hospital, Rouen, . Dr D. Maltête, Pr. D. Hannequin, Dr. O. Martinaud, Dr E. Gérardin, Pr. B. Mihout, Mmes C. Aubier-Girard, S Bioux, E. Bliaux, D. Pouliquen

Caen :

- Department of Neurology, University Hospital,Caen, : Pr G. Defer, Pr F. Viader, Dr Guillamo Dr Marié, Dr Carluer, Mme Lebrun

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of Parkinson's disease: Gibb and Gelb criteria
* Apathy defined by a score of - 16 or more on the LARS scale (Sockeel et al., 2006)and criteria of Marin (1991)
* No dementia according to DSM IV with MMSE Score≥ 27 and Mattis score≥ 130
* Under stable dopaminergic treatment for 3 months

Exclusion criteria:

* Depression according to DSM-IV criteria and a score < 18 on the MADRS
* Subthalamic stimulation of less than one year
* Subthalamic stimulation without stable parameters for 3 months
* Subject older than 80 years
* Severe rest tremor with a subscore > or= 3 on the UPDRS part
* Parkinson related Psychosis in progress
* Hypersensibility to cholinesterase inhibitors or carbamates
* Myocardial infarction, other cardiac affections
* Severe hepatic insufficiency
* Sever medical illness
* Skin diseases interfering with transdermal patch
* Pregnancy
* Incapacity to give the consent

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Measure on the scale : Lille Apathy Rating Scale (LARS) | 6 months
  measure of the reduction of apathy with this qualitative scale from -36 +36 with the cut off -16

SECONDARY OUTCOMES:
Cognitive, motor and behaviour assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Principal Investigator — Department of Neurology, University Hospital, Lille
Locations (1):
- Devos, Lille, Nord, France

REFERENCES:
- [Derived] Devos D, Moreau C, Maltete D, Lefaucheur R, Kreisler A, Eusebio A, Defer G, Ouk T, Azulay JP, Krystkowiak P, Witjas T, Delliaux M, Destee A, Duhamel A, Bordet R, Defebvre L, Dujardin K. Rivastigmine in apathetic but dementia and depression-free patients with Parkinson's disease: a double-blind, placebo-controlled, randomised clinical trial. J Neurol Neurosurg Psychiatry. 2014 Jun;85(6):668-74. doi: 10.1136/jnnp-2013-306439. Epub 2013 Nov 11. PMID 24218528